CLINICAL TRIAL: NCT04083846
Title: A Randomized, Open-label, Single Dose, Crossover Study to Investigate the Pharmacokinetic Profiles and Safety of High-dose CKD-385 in Healthy Volunteers Under Fed Conditions
Brief Title: Clinical Study to Investigate the Pharmacokinetic Profiles and Safety of High-dose CKD-385 in Healthy Volunteers(Fed)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A88_04BE1911P
Record Dates: First submitted 2019-09-08; First posted 2019-09-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): 1. Period 1: Reference drug
  2. Period 2: Test drug 1
  3. Period 3: Test drug 2
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 2 (Experimental): 1. Period 1: Test drug 2
  2. Period 2: Reference drug
  3. Period 3: Test drug 1
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 3 (Experimental): 1. Period 1: Test drug 1
  2. Period 2: Test drug 2
  3. Period 3: Reference drug
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 4 (Experimental): 1. Period 1: Test drug 2
  2. Period 2: Test drug 1
  3. Period 3: Reference drug
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 5 (Experimental): 1. Period 1: Test drug 1
  2. Period 2: Reference drug
  3. Period 3: Test drug 2
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2
- Group 6 (Experimental): 1. Period 1: Reference drug
  2. Period 2: Test drug 2
  3. Period 3: Test drug 1
  Interventions: Drug: Reference drug; Drug: Test drug 1; Drug: Test drug 2

INTERVENTIONS:
Drug: Reference drug — D744 Cap. 1 Cap., single oral administration under fed condition
  Other Names: D744
Drug: Test drug 1 — CKD-385 64 mg formulation I Tab. 1 Tab., single oral administration under fed condition
  Other Names: CKD-385 64 mg formulation I
Drug: Test drug 2 — CKD-385 64 mg formulation II Tab. 1 Tab., single oral administration under fed condition
  Other Names: CKD-385 64 mg formulation II

SUMMARY:
This study is a randomized, open-label, fed, single dose, crossover study to investigate the pharmacokinetic profiles and safety of high-dose CKD-385 in healthy volunteers under fed conditions.

DETAILED DESCRIPTION:
To healthy subjects of twenty-four (24), following treatments are administered dosing in each period and wash-out period is a minimum of 7 days. Reference drug: D744, Test drug 1: CKD-385 64 mg formulation I, Test drug 2: CKD-385 64 mg formulation II. Pharmacokinetic blood samples are collected up to 48 hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria

1. Healthy adult aged over 19 at the time of screening
2. Subject who had 17.5kg/m² ≤ Body Mass Index (BMI) < 30.5kg/m² and a total body weight ≥ 55 kg

   # BMI=Weight(kg) / Height(m)²
3. Subject without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years
4. Subject who were deemed to be appropriate as study subjects in accordance with the screening results (laboratory tests, vital signs, ECG etc.)
5. Subject who signed an informed consent form approved by the Institutional Review Board(IRB) of Chonbuk National University Hospital and decided to participate in the study after being fully informed of the study prior to participation, including the objective, content and characteristics of the investigational drug
6. Subject who must consent to the use of reliable contraception and not to donate sperm, from the 1st administration of the investigational product until 1 month after the last administration of investigational product
7. Subject with the ability and willingness to participate during the study period

Exclusion Criteria

1. Subject who has medical evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, urinary, cardiovascular, hepatic, psychiatric, neurologic or allergic diseases
2. Subject with a medical history of gastrointestinal disorders(esophageal achalasia or esophagus stenosis, Crohn's disease) or gastrointestinal surgery(except for simple appendicitis surgery or hernia surgery or tooth extraction surgery) that may affect the absorption of drug
3. Subject who shows the following values as a result of laboratory tests

   *Alanine Transaminase(ALT) or Aspartate Transaminase(AST) > 2 times upper limit of normal range
4. Subject who has a history of regular alcohol consumption in excess of 210 g/week within 6 months prior to screening
5. Subject who smokes more than 20 cigarettes a day within 6 months prior to screening
6. Subject who took other clinical trial drugs or bioequivalence test drugs within 6 months before the first administration of clinical trial drug
7. Subject who conform to the specific items below

   * systolic blood pressure less than 90 mmHg, not less than 140 mmHg or diastolic blood pressure less than 60 mmHg or not less than 90 mmHg in a sitting position
   * Severe bradycardia (less than 50 beats/minute)
8. Subject who has a medical history of significant alcohol abuse or drug abuse within one year prior to screening
9. Subject who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first administration of investigational product(s).
10. Subject who uses any of other drugs, including over-the-counter medications and prescription medications within 10 days prior to first administration of investigational product(s).
11. Subject who donated whole blood within 2 months, or blood components within 1 month prior to first administration of investigational product(s).
12. Subject who has hypersensitivity to investigational product(s) or investigational product(s) ingredient.
13. Subject is unable to consume a high-fat meal provided during the study.
14. Subject who were deemed to be inappropriate to participate in the study by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Area Under Curve last(AUCt) | Pre-dose (0 hour), post-dose 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  Area under the plasma concentration time curve of CKD-385 64 mg formulation Ⅰ/D744 or CKD-385 64 mg formulation Ⅱ/D744, from time zero up to the last measurable concentration.
Cmax | Pre-dose (0 hour), post-dose 1, 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48 hours
  The maximum concentration observed of CKD-385 64 mg formulation Ⅰ/D744 or CKD-385 64 mg formulation Ⅱ/D744 over blood sampling time.

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No